CLINICAL TRIAL: NCT04827966
Title: A Randomized Controlled Trial on the Remineralization Agents Used for the Treatment of White Spot Lesions
Brief Title: Remineralization Agents for the Treatment of White Spot Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Ministry of Health, Bahrain (Other Government)
Responsible Party: Principal Investigator, Gowri Sivaramakrishnan, Specialist Prosthodontist and Dental Tutor, Ministry of Health, Bahrain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOHWS
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: White Spot Lesion of Tooth
Keywords: fluoride; remineralization; esthetics; orthodontic brackets
MeSH Terms: interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Fluoride Varnish (Active Comparator): Clinpro® is 5% sodium fluoride varnish and is indicated to be used for hypersensitive as well as for demineralized teeth. It flows smoothly on moist teeth and binds firmly to their surfaces. 1ml of Clinpro® contain 50 mg of sodium fluoride. 0.2-0.5ml of the varnish is applied onto the tooth surface after through cleaning. One coats of the varnish will be applied and patient will be instructed not to rinse with water or eat for 30 minutes. This is based on the manufacturer's instructions.
  Interventions: Other: Clinpro® 5% sodium fluoride plus tri calcium phosphate varnish
- Tooth Mousse (Active Comparator): Tooth Mousse® contains Casein phosphopeptide-Amorphous calcium phosphate (CPP - ACP) is product from the milk casein. This delivers the necessary Calcium and Phosphate ions to the tooth, which will reduce the risk of caries and white spot by enhancing tooth remineralization. One tube of the Tooth Mousse will be prescribed to the patient. Patient will be instructed to apply the product using finger every night after brushing and flossing. This is continued till the prescribed product is finished. This is approximately calculated to be about 8 to 12 weeks.Patient is instructed to leave the paste for about 3 minutes and then rinse. This is based on the manufacturer's instructions.
  Interventions: Other: Tooth Mousse® - Casein phosphopeptide-Amorphous calcium phosphate (CPP - ACP)s
- MI Paste (Active Comparator): MI Paste® which is Casein phosphopeptide-Amorphous calcium phosphate fluoride (CPP-ACPF) additional contains fluoride in addition to CPP-ACP. The level of fluoride is 900ppm which approximates that in adult strength toothpastes. Recent studies have investigated the remineralization potential of CPP-ACP combined with fluoride and have found a synergistic effect when these are administered together, which is the composition in MI paste. One tube of the MI Paste will be prescribed to the patient. Patient will be instructed to apply the product using finger every night after brushing and flossing. This is continued till the prescribed product is finished. This is approximately calculated to be about 8 to 12 weeks.Patient is instructed to leave the paste for about 3 minutes and then rinse. This is based on the manufacturer's instructions.
  Interventions: Other: MI Paste® -Casein phosphopeptide-Amorphous calcium phosphate fluoride (CPP-ACPF)
- Acidulated phosphate fluoride gel (Active Comparator): A stable thixotropic gel providing 1.23% fluoride ion. This is only for professional use and applied by the dentist. The teeth is cleaned and polished and the gel is applied onto a tray. It is filled upto one third of the tray according to manufacturer's instructions. The tray is then inserted into the mouth and the patient is asked to gently bite down lightly for 1 to 4 minutes.The tray is then removed and patient is asked to expectorate any material in the mouth. The patient is instructed not to eat, rinse or drink for 30 minutes.
  Interventions: Other: Zap® 1.23% APF gel - Acidulated phosphate fluoride
- Fluoride Mouthrinse (Active Comparator): Listerine® Sodium fluoride (0.2%) mouth rinses are effective in reducing caries and inhibit carbohydrate utilization of oral microorganisms by blocking enzymes involved in the bacterial glycolytic pathway studies have shown sodium fluoride mouth rinse to be effective in reducing S. mutans counts.
  Interventions: Other: Listerine fluoride mouthrinse

INTERVENTIONS:
Other: Clinpro® 5% sodium fluoride plus tri calcium phosphate varnish — Clinpro® is 5% sodium fluoride varnish and is indicated to be used for hypersensitive as well as for demineralized teeth. It flows smoothly on moist teeth and binds firmly to their surfaces. 1ml of Clinpro® contain 50 mg of sodium fluoride
  Arms: Fluoride Varnish
Other: Tooth Mousse® - Casein phosphopeptide-Amorphous calcium phosphate (CPP - ACP)s — Tooth Mousse® contains Casein phosphopeptide-Amorphous calcium phosphate (CPP - ACP) is product from the milk casein. This delivers the necessary Calcium and Phosphate ions to the tooth, which will reduce the risk of caries and white spot by enhancing tooth remineralization.
  Arms: Tooth Mousse
Other: MI Paste® -Casein phosphopeptide-Amorphous calcium phosphate fluoride (CPP-ACPF) — MI Paste® which is Casein phosphopeptide-Amorphous calcium phosphate fluoride (CPP-ACPF) additional contains fluoride in addition to CPP-ACP. The level of fluoride is 900ppm which approximates that in adult strength toothpastes.
  Arms: MI Paste
Other: Zap® 1.23% APF gel - Acidulated phosphate fluoride — 1.23% APF (Acidulated phosphate fluoride) gel is routinely used professional based fluoride for patients with high caries risk.
  Arms: Acidulated phosphate fluoride gel
Other: Listerine fluoride mouthrinse — Listerine® Sodium fluoride (0.2%) mouth rinses are effective in reducing caries and inhibit carbohydrate utilization of oral microorganisms by blocking enzymes involved in the bacterial glycolytic pathway studies have shown sodium fluoride mouth rinse to be effective in reducing S. mutans counts
  Arms: Fluoride Mouthrinse

SUMMARY:
Clinically, formation of white spots can occur as early as 4 weeks into orthodontic treatment and very common in high caries risk individuals. When left untreated, the calcium loss continues, the enamel breaks down entirely, and a cavity appears. These can cause caries thereby leading to poor esthetics and patient dissatisfaction. The labio-gingival area of the lateral incisors is the most common site for WSL and the maxillary posterior segments are the least common site, with males affected more in comparison with females.Hence inducing remineralization of existing lesions is the key treatment to prevent cavitation.

DETAILED DESCRIPTION:
White spot lesion (WSL) is the earliest sign of demineralization of the enamel and a common problem caused because of plaque accumulation and poor oral hygiene. These WSLs are of great concern in young patients, considering that esthetics is the prime reason for young patients to seek dental treatment. The appearance of these areas of demineralization should be prevented and appropriate strategies must be undertaken in remineralizing these lesions. A recent meta-analysis on the incidence and prevalence of these lesions in orthodontic patients included 14 studies indicated that the incidence of new carious lesions formed during orthodontic treatment in patients was 45.8% and the prevalence of lesions in patients undergoing orthodontic treatment was 68.4%. This is considerably high and needs urgent attention.

Enamel decalcification can occur as a result of orthodontic bracket or any other foreign body attached onto the tooth surface, and provoked by poor oral hygiene. It is an incipient caries in the subsurface beneath an intact enamel outer surface. It is characterized by chalky white appearance (WSLs) mostly around the brackets, and have different refractive index than intact enamel surface.If the WSL's are left untreated it can progress to break down the enamel surface and develop into advance stages of carious lesion that indicate esthetic restorations or in more advance cases a prosthodontic intervention.

Research has shown good evidence on non-invasive treatment of WSLs such as establishing good oral hygiene and the use of fluoride and non-fluoride remineralizing agents. Fluoride containing agents are available as high-fluoride toothpaste, fluoride mouthwash, gels and varnish. Recently, other non-fluoride materials and techniques such as casein phosphopeptide -amorphous calcium phosphate (CPP-ACP) has shown promising results.

Clinpro® is 5% sodium fluoride varnish and is indicated to be used for hypersensitive as well as for demineralized teeth. It flows smoothly on moist teeth and binds firmly to their surfaces. 1ml of Clinpro® contain 50 mg of sodium fluoride. Fluoride varnish placed around orthodontic brackets during treatment has been shown to reduce the incidence and prevalence of WSL. Tooth Mousse® contains Casein phosphopeptide-Amorphous calcium phosphate (CPP - ACP) is product from the milk casein. This delivers the necessary Calcium and Phosphate ions to the tooth, which will reduce the risk of caries and white spot by enhancing tooth remineralization. MI Paste® which is Casein phosphopeptide-Amorphous calcium phosphate fluoride (CPP-ACPF) additional contains fluoride in addition to CPP-ACP. The level of fluoride is 900ppm which approximates that in adult strength toothpastes. When CPP-ACPF is applied in the oral environment, it will bind to biofilms, plaque, bacteria, hydroxyapatite and soft tissue localizing bio-available calcium, phosphate and fluoride. Recent studies have investigated the remineralization potential of CPP-ACP combined with fluoride and have found a synergistic effect when these are administered together, which is the composition in MI paste. Patients who have previous history of milk protein allergy or lactose intolerance are not suitable to use MI paste or tooth mousse. This is based on the manufacturer's instructions. However, there is no published data on these allergic reactions to CPP-ACP products so far. 1.23% APF (Acidulated phosphate fluoride) gel is routinely used professional based fluoride for patients with high caries risk. Listerine® Sodium fluoride (0.2%) mouth rinses are effective in reducing caries and inhibit carbohydrate utilization of oral microorganisms by blocking enzymes involved in the bacterial glycolytic pathway studies have shown sodium fluoride mouth rinse to be effective in reducing S. mutans counts.

Considering the variety of agents that are available the aim of this clinical study is to compare Clinpro® 5% sodium fluoride plus tri calcium phosphate varnish, Tooth mousse® CPP-ACP without fluoride, MI Paste® CPP-ACP with fluoride and 0.2% sodium fluoride mouthwash in remineralization of white spot lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending the dental clinic for treatment of white spot lesions on their teeth
* using fluoride toothpaste once or twice daily for brushing
* does not use any other form of fluoride
* history of recent fixed orthodontic treatment
* presenting with white spot lesions on minimum of three anterior or posterior teeth on the labial surfaces
* provide written informed consent

Exclusion Criteria:

* Patients who do not fit into the above mentioned inclusion criteria.
* Patients who are allergic to milk or any other milk products will be excluded from the study. Milk protein allergy and lactose intolerance tests will be performed on participants belonging to active comparators Tooth Mousse and MI paste which contain casein phosphoprotein before enrolling them in the trial.
* Patients who are vegan and do not use or consume any animal products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Enamel decalcification score recorded using Enamel decalcification index (EDI) by Banker and Richmond | Baseline (before treatment)
  The index is used to score the demineralisation of 4 tooth surfaces- mesial, distal, incisal and gingival.
Enamel decalcification score recorded using Enamel decalcification index (EDI) by Banker and Richmond | 3 weeks following treatment
  The index is used to score the demineralisation of 4 tooth surfaces- mesial, distal, incisal and gingival.
Enamel decalcification score recorded using Enamel decalcification index (EDI) by Banker and Richmond | 6 weeks following treatment
  The index is used to score the demineralisation of 4 tooth surfaces- mesial, distal, incisal and gingival.
Enamel decalcification score recorded using Enamel decalcification index (EDI) by Banker and Richmond | 9 weeks following treatment
  The index is used to score the demineralisation of 4 tooth surfaces- mesial, distal, incisal and gingival.

SECONDARY OUTCOMES:
Number of patients with any adverse effects | 3 weeks
  Any adverse effects reported in the form of allergy , hypersensitivity, discoloration.
Number of patients with any adverse effects | 6 weeks
  Any adverse effects reported in the form of allergy , hypersensitivity, discoloration.
Number of patients with any adverse effects | 9 weeks
  Any adverse effects reported in the form of allergy , hypersensitivity, discoloration.

CONTACTS AND LOCATIONS:
Locations (1):
- Halet bu maher health center, Al Muharraq, Bahrain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umeh OD, Utomi IL, Ndukwe AN, Izuka M. Demineralization preventive practices among Nigerian orthodontists-An evidence-based approach? Niger J Clin Pract. 2020 May;23(5):589-595. doi: 10.4103/njcp.njcp_315_19. PMID 32367863
- [Background] Memarpour M, Shafiei F, Rafiee A, Soltani M, Dashti MH. Effect of hydroxyapatite nanoparticles on enamel remineralization and estimation of fissure sealant bond strength to remineralized tooth surfaces: an in vitro study. BMC Oral Health. 2019 May 28;19(1):92. doi: 10.1186/s12903-019-0785-6. PMID 31138191
- [Result] Goswami M, Saha S, Chaitra TR. Latest developments in non-fluoridated remineralizing technologies. J Indian Soc Pedod Prev Dent. 2012 Jan-Mar;30(1):2-6. doi: 10.4103/0970-4388.95561. PMID 22565510
- [Result] Pradeep K, Kumar PR. Remineralizing agents in the non-invasive treatment of early carious lesions. Int J Dent Case Rep 2011; 1:73-84.
- [Result] Sonesson M, Bergstrand F, Gizani S, Twetman S. Management of post-orthodontic white spot lesions: an updated systematic review. Eur J Orthod. 2017 Apr 1;39(2):116-121. doi: 10.1093/ejo/cjw023. PMID 27030284
- [Result] Fernandez-Ferrer L, Vicente-Ruiz M, Garcia-Sanz V, Montiel-Company JM, Paredes-Gallardo V, Almerich-Silla JM, Bellot-Arcis C. Enamel remineralization therapies for treating postorthodontic white-spot lesions: A systematic review. J Am Dent Assoc. 2018 Sep;149(9):778-786.e2. doi: 10.1016/j.adaj.2018.05.010. Epub 2018 Jul 12. PMID 30007454
- [Result] Khoroushi M, Kachuie M. Prevention and Treatment of White Spot Lesions in Orthodontic Patients. Contemp Clin Dent. 2017 Jan-Mar;8(1):11-19. doi: 10.4103/ccd.ccd_216_17. PMID 28566845
- [Result] Cosma LL, Suhani RD, Mesaros A, Badea ME. Current treatment modalities of orthodontically induced white spot lesions and their outcome - a literature review. Med Pharm Rep. 2019 Jan;92(1):25-30. doi: 10.15386/cjmed-1090. Epub 2019 Jan 15. PMID 30957083